CLINICAL TRIAL: NCT07186387
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Study to Evaluate the Efficacy, Safety, and Tolerability of LW402 in Patients With Moderate-to-Severe Atopic Dermatitis
Brief Title: Study of LW402 in Moderate-to-Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Longwood Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LW402-II-02
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2023-05

CONDITIONS: Atopic Dermatitis (AD)
Keywords: Moderate-to-severe
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LW402 Low Dose (Experimental): LW402 administered orally, BID (low dose)
  Interventions: Drug: LW402
- LW402 Medium Dose (Experimental): LW402 administered orally, BID (medium dose)
  Interventions: Drug: LW402
- LW402 High Dose (Experimental): LW402 administered orally, BID (high dose)
  Interventions: Drug: LW402
- Placebo (Placebo Comparator): LW402 placebo administered orally, BID
  Interventions: Drug: LW402 placebo

INTERVENTIONS:
Drug: LW402 — LW402 tablets
  Arms: LW402 High Dose; LW402 Low Dose; LW402 Medium Dose
Drug: LW402 placebo — LW402 placebo tablets
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double blind, placebo-controlled phase 2 study to evaluate the efficacy, safety, PK and PD ofLW402 in patients with moderate-to-severe atopic dermatitis.

DETAILED DESCRIPTION:
The study consists of an up-to-4-week screening period, a 12-week double-blind treatment period and a 4-week safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with AD for at least 12 months before Screening, with below requirements: 1) EASI score ≥16 at Screening and Baseline; 2) IGA score ≥3 at Screening and Baseline; 3) ≥10% BSA of AD involvement at Screening and Baseline

Exclusion Criteria:

* Not enough washing-out period for previous therapy. Concurrent disease/status which may potentially affect the efficacy/safety judgement.

pregnancy. Other.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2023-05-11 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
Proportion of participants achieving EASI-50 at week 12 | 12 weeks
  Proportion of participants achieving EASI-50 (≥50% reduction from baseline in Eczema Area and Severity Index score) at week 12.
  The EASI is a composite index with scores ranging from 0 to 72. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) will each be assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe).

SECONDARY OUTCOMES:
Proportion of participants achieving EASI-75 at week 12 | 12 weeks
  Proportion of participants achieving EASI-75 (≥75% reduction from baseline in Eczema Area and Severity Index score) at week 12.
Proportion of participants with IGA score of 0 or 1 and a reduction of IGA score by ≥2 points from baseline at week 12 | 12 weeks
  Proportion of participants with Investigator's Global Assessment (IGA) score of 0 or 1 and a reduction of IGA score by ≥2 points from baseline at week 16.
  IGA is an assessment instrument used in clinical studies to rate the severity of AD globally, based on a 6-point scale ranging from 0 (clear) to 5 (very severe).
Incidence of adverse events (AEs), abnormal physical examinations, abnormal vital signs, abnormal ECG, and abnormal lab testing. | 16 weeks
  Incidence of adverse events (AEs), abnormal physical examinations, abnormal vital signs, abnormal ECG, and abnormal lab testing.
PD: pSTAT3 and pSTAT5 inhibition rates | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No